CLINICAL TRIAL: NCT04263441
Title: Navigating Insurance Coverage Expansion (NICE): A Collaboration to Increase Access to Care for Black and Hispanic Men Who Have Sex With Men and Transgender Persons
Brief Title: Navigating Insurance Coverage Expansion (NICE)
Acronym: NICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Howard Brown Health Center (Other); Chicago House and Social Service Agency (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB16-1260; CDC (Other Grant/Funding Number: RFA-PS-16-004)
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: HIV/AIDS
Keywords: Pre-Exposure Prophylaxis (PrEP)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NICE Intervention (Experimental): The proposed intervention will engage clients in the health care enrollment and navigation process in-person, at the time of the HIV testing event. Subjects will be asked to share thoughts on the satisfaction survey.
  Interventions: Behavioral: NICE Intervention
- Control Intervention (No Intervention): Subjects will be offered a handout on how to enroll in healthcare coverage This group will be provided with the site's standard healthcare enrollment and linkage to care, which is specific to the health care clinic they are visiting. Subjects will be followed for 1 year and information including lab tests and insurance coverage status will be collected. This information will be collected from medical record review. Subjects will be asked to share thoughts on the satisfaction survey.

INTERVENTIONS:
Behavioral: NICE Intervention — Subjects enrolled in the intervention arm will be offered assistance in enrolling in healthcare coverage and provided assistance on where they can go for care immediately. Subjects will be followed for 1 year and information including lab tests and insurance coverage status will be collected. This information will be collected from medical record review.
  Arms: NICE Intervention

SUMMARY:
The purpose of this research is to measure the effectiveness of an in-person assistance intervention on successful insurance enrollment, types of insurance coverage, rates of linkage to and retention in HIV-related health care, referrals to other HIV-associated health services, and health outcomes. The study population is Black and Hispanic men who have sex with men (MSM) and transgender persons who are at higher risk for HIV.

The study team will be testing the hypotheses that in-person health insurance enrollment assistance results in positive outcomes with regard to linkage to and retention in HIV-related health care. Analyses will be used to assess the efficacy of the intervention as an emerging practice.

DETAILED DESCRIPTION:
The overall goal of this study is to test whether providing in-person assistance in enrolling in private health insurance or Medicaid for the first time, changing to a different insurance plan, or understanding how to use current insurance policies following HIV testing will (1) increase the proportion of participants who obtain health insurance; (2) result in better health outcomes among participants; (3) improve the linkage and retention rates of participants, especially those diagnosed with HIV; and (4) increase linkage and retention rates sufficiently to justify the cost of implementing the intervention (cost-benefit analysis).

ELIGIBILITY:
Inclusion Criteria:

* Black or Hispanic men who have sex with men (MSM) or transgender persons
* 18 or older

Exclusion Criteria:

* Cisgender women
* Cisgender men who have not had anal or oral sex with a man in last 2 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Linkage | 30 days
  Proportion of participants who completed at least one HIV-related medical visit within 30 days after their baseline HIV test was performed
Delayed Linkage | 90 days
  Proportion of participants who completed at least one HIV-related medical visit within 90 days after their baseline HIV test was performed
Retention | 365 days
  Proportion of HIV positive participants who completed at least 2 HIV-related medical visits within 12 months after their baseline HIV test was performed. Visits must be separated by at least 3 months.
Early Retention | 183 days
  Proportion of HIV negative participants who completed at least 2 medical visits within 6 months after their baseline HIV test was performed, regardless of whether they enrolled in PrEP.

SECONDARY OUTCOMES:
Linkage | 365 Days
  Median length of time between baseline HIV test and first completed HIV-related care visit
Retention | 365 Days
  Median length of time between first completed HIV-related care visit and subsequent HIV-related care visits during the 12-month follow-up period
Viral Load Reduction | 91 days
  Proportion of HIV positive participants who are retained and achieved reduced viral load at their first visit at least 3 months post-linkage. Reduced viral load is considered to be fewer RNA copies/mL than the participant's viral load test result on their previous medical care visit.
Viral Suppression | 365 days
  Proportion of HIV positive participants who are retained and achieved viral suppression (<200 RNA copies/mL) at their last visit within 12 months after enrollment
Maintained Status | 365 days
  Proportion of HIV negative participants who are retained and remained HIV negative at their last visit within 12 months after enrollment, regardless of whether they enrolled in PrEP.
Enrolled in Insurance | At study enrollment
  Proportion of intervention arm participants who are successfully enrolled in health insurance
Changed Insurance | At study enrollment
  Proportion of currently insured intervention arm participants who change their insurance plan and reasons why
Medicaid Enrollment | At study enrollment
  Proportion of newly enrolled intervention arm participants who enroll in Medicaid
Private Insurance Enrollment | At study enrollment
  Proportion of newly enrolled intervention arm participants who enroll in private health insurance
Market place enrollment | At study enrollment
  Proportion of intervention arm participants who enroll in the bronze level of coverage, who enroll in the silver level of coverage, and who enroll in gold or platinum levels of coverage

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Howard Brown Health, Chicago, Illinois
  - Chicago House and Social Service Agency, Inc., Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herbst JH, Jacobs ED, Finlayson TJ, McKleroy VS, Neumann MS, Crepaz N; HIV/AIDS Prevention Research Synthesis Team. Estimating HIV prevalence and risk behaviors of transgender persons in the United States: a systematic review. AIDS Behav. 2008 Jan;12(1):1-17. doi: 10.1007/s10461-007-9299-3. Epub 2007 Aug 13. PMID 17694429
- [Background] Millett GA, Peterson JL, Flores SA, Hart TA, Jeffries WL 4th, Wilson PA, Rourke SB, Heilig CM, Elford J, Fenton KA, Remis RS. Comparisons of disparities and risks of HIV infection in black and other men who have sex with men in Canada, UK, and USA: a meta-analysis. Lancet. 2012 Jul 28;380(9839):341-8. doi: 10.1016/S0140-6736(12)60899-X. Epub 2012 Jul 20. PMID 22819656
- [Background] Sullivan PS, Rosenberg ES, Sanchez TH, Kelley CF, Luisi N, Cooper HL, Diclemente RJ, Wingood GM, Frew PM, Salazar LF, Del Rio C, Mulligan MJ, Peterson JL. Explaining racial disparities in HIV incidence in black and white men who have sex with men in Atlanta, GA: a prospective observational cohort study. Ann Epidemiol. 2015 Jun;25(6):445-54. doi: 10.1016/j.annepidem.2015.03.006. Epub 2015 Mar 24. PMID 25911980
- [Background] Khan L. Transgender health at the crossroads: legal norms, insurance markets, and the threat of healthcare reform. Yale J Health Policy Law Ethics. 2011 Summer;11(2):375-418. No abstract available. PMID 22136012
- [Background] Hall G, Li K, Wilton L, Wheeler D, Fogel J, Wang L, Koblin B. A Comparison of Referred Sexual Partners to Their Community Recruited Counterparts in The BROTHERS Project (HPTN 061). AIDS Behav. 2015 Dec;19(12):2214-23. doi: 10.1007/s10461-015-1005-2. PMID 25874753
- [Background] Matts JP, Lachin JM. Properties of permuted-block randomization in clinical trials. Control Clin Trials. 1988 Dec;9(4):327-44. doi: 10.1016/0197-2456(88)90047-5. PMID 3203524
- [Background] Farnham PG, Sansom SL, Hutchinson AB. How much should we pay for a new HIV diagnosis? A mathematical model of HIV screening in US clinical settings. Med Decis Making. 2012 May-Jun;32(3):459-69. doi: 10.1177/0272989X11431609. Epub 2012 Jan 12. PMID 22247422
- [Background] Gebo KA, Fleishman JA, Conviser R, Hellinger J, Hellinger FJ, Josephs JS, Keiser P, Gaist P, Moore RD; HIV Research Network. Contemporary costs of HIV healthcare in the HAART era. AIDS. 2010 Nov 13;24(17):2705-15. doi: 10.1097/QAD.0b013e32833f3c14. PMID 20859193
- [Background] Horberg M, Raymond B. Financial policy issues for HIV pre-exposure prophylaxis: cost and access to insurance. Am J Prev Med. 2013 Jan;44(1 Suppl 2):S125-8. doi: 10.1016/j.amepre.2012.09.039. No abstract available. PMID 23253752
- See also: The 10 largest Hispanic origin groups: Characteristics, rankings, top Counties — https://www.pewresearch.org/hispanic/2012/06/27/the-10-largest-hispanic-origin-groups-characteristics-rankings-top-counties/
- See also: Injustice at Every Turn: A Report of the National Transgender Discrimination Survey — https://www.thetaskforce.org/wp-content/uploads/2019/07/ntds_full.pdf
- See also: Moving Black MSM Along the HIV Care Continuum — https://files.hiv.gov/s3fs-public/bmsm-webinar-06252014.pdf
- See also: In-Person Assistance in the Health Insurance Marketplaces — http://www.cms.gov/cciio/programs-and-initiatives/health-insurance-marketplaces/assistance.html
- See also: Chicago Department of Public Health. HIV/STI Surveillance Report 2016 — https://www.chicago.gov/content/dam/city/depts/cdph/HIV_STI/World_AIDS_Day_Report_012717.pdf
- See also: HIV Risk and Prevention Behaviors Among Men Who Have Sex With Men, Chicago, 2008 and 2011 — https://www.chicago.gov/content/dam/city/depts/cdph/infectious_disease/STI_HIV_AIDS/MSMReport2012.pdf